CLINICAL TRIAL: NCT03518450
Title: Early Mobilization and Postoperative Analgesia After Total Knee Arthroplasty, a Prospective Comparative Study: Adductor Canal Block vs. Femoral Nerve Block vs. Apex Femoral Triangle Block
Brief Title: Femoral Triangle Block: Early Mobilization and Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)299/2017
Record Dates: First submitted 2018-03-17; First posted 2018-05-08 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-11

CONDITIONS: Arthroplasty, Replacement, Knee; Anesthesia, Conduction; Pain, Postoperative; Ultrasonography, Interventional
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Femoral Nerve Block (Active Comparator): Ultrasound guided femoral nerve block, 30 ml of 0.25% bupivacaine and 4 mg of dexamethasone to be administered.
  Interventions: Procedure: Femoral Nerve Block
- Adductor Canal Block (Active Comparator): Ultrasound guided adductor canal block, at the proximal third of the canal, 30 ml of 0.25% bupivacaine and 4 mg of dexamethasone to be administered.
  Interventions: Procedure: Adductor Canal Block
- Apex Femoral Triangle Block (Experimental): Ultrasound guided femoral triangle block, at the distal third of the triangle, 30 ml of 0.25% bupivacaine and 4 mg of dexamethasone to be administered.
  Interventions: Procedure: Apex Femoral Triangle Block

INTERVENTIONS:
Procedure: Apex Femoral Triangle Block — Nerve block that aims the vastus medialis nerve, the saphenous nerve and the anterior femoral cutaneous nerve.
  Arms: Apex Femoral Triangle Block
Procedure: Femoral Nerve Block — Regional anesthetic technique that blocks the sensory and motor information of the femoral nerve (and it's branches).
  Arms: Femoral Nerve Block
Procedure: Adductor Canal Block — Interfascial block that targets mainly the saphenous nerve.
  Arms: Adductor Canal Block

SUMMARY:
The objective of this trial is to compare the efficacy of three different nerve blocks as an analgesic option after total knee arthroplasty (TKA), based on muscle strength, mobilization and pain.

The Adductor Canal Block has been proposed as an equally effective technique to the Femoral Nerve Block in terms of pain control after a TKA, with the benefit of preserving muscle function. We hypothesize that a block performed at the apex of the femoral triangle would best balance analgesia with quadriceps function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any gender, from 18 to 90 years old that accept to participate in the study.
* Programmed primary total knee arthroplasty surgery

Exclusion Criteria:

* Emergent surgery
* Reinterventions
* Unstable psychiatric pathology, dementia
* Kidney or hepatic disease that contraindicates the use of NSAIDs and/or Paracetamol.
* Allergy to amides local anesthesics, NSAIDs, opioids and/or Paracetamol.
* Daily use of opioids greater than 30 mg of morphine (or equivalent)
* Patients under 18 or over 90 years old.
* Drug abuse
* Rejection to be a participant of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Maximum voluntary isometric contraction (MVIC) | 6 hours postoperatively
  It measures quadriceps strength and is normalized to the body mass index (N * m/kg). This test correlates well with the functional outcome. Will be measured with standard handheld dynamometer (MicroFET2; Hoogan Industries, West Jordan, Utah) perpendicular to the tibial crest 5 cm proximal to the medial malleolus to make the measurement. The patients are told to "reach maximum force and hold for three seconds." Three measurements will be done, and the average will be taken.
  The primary effectiveness endpoints of the study will be the percentage of baselineMVIC retained on the quadriceps of the leg receiving arthroplasty for each subject at 6 hours postoperatively.
  A higher the percentage will relate with less motor block.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | 6, 24 and 48 hours postoperatively.
  Timed Up and Go gauges a patient's sense of balance by measuring the time required for a certain set of movements: stand up from a chair, walk 3 m, walk back, and sit down. It has been verified to serve as a good indicator of functional level.
  Measured in seconds, the better values are related to shorter times.
30' CST (30 secs Chair Stand Test) | 6, 24 and 48 hours postoperatively.
  How many times can a patient stand up and sit down from a chair in 30 seconds. The amount of times will be counted, more times will be related to a better outcome.
Range of Motion (ROM) | 6, 24 and 48 hours postoperatively.
  Range of motion refers to a knee's degree of extension or flexion and is measured via a goniometer. Considering normal values from 0-120º, the baseline movement will be measured preoperatively to be compared postoperatively.
Daniels' Test | 6, 24 and 48 hours postoperatively.
  Active extension of the knee against gravity and applied resistance (0-5). 5: normal contraction against gravity and maximal resistance. 0: abscence of contraction.
10-PMS (10 point Mobility Scale) | 6, 24 and 48 hours postoperatively.
  Scale from 0-10 in which the mobility of the patient is measured; sitting on the bed, chair, edge of the bed, mobilize the knee more than 45º, stand up, walk with or without a mobility aid.
  Higher values are related to better outcomes.
  An expected degree of flexion of the knee is ≥45 degrees on postoperative day 1 and ≥70 degrees on postoperative day 3.
  Expected points for postoperative day 0: 4 points Expected points for postoperative day 1: 8 points Expected points for postoperative day 2: 9-10 points
Pain measurement trough the visual analogue scale (VAS) | 6, 24 and 48 hours postoperatively.
  Pain will be measured via the VAS pain score by having the patient point on an unmarked scale how their pain was and then translating it to millimeters on the 100-mm scale.
  0 mm: no pain 100 mm: severe/extreme pain
Quantity of opioids administered | 6, 24 and 48 hours postoperatively.
  into morphine equivalent if needed.
APS-POQ-R. | At 24 hours postoperatively
  Developed by an interdisciplinary task force of members of the American Pain Society, the Patient Outcome Questionnaire (APS-POQ) for QI has been revised to include instrument psychometrics. The article is available by open access at The Journal of Pain web site.
Patient satisfaction | 24 and 48 hours postoperatively
  Scale from 0 to 10, answering how do they feel about the treatment received, being 10 the maximum value related to the highest satisfaction level.
Length of hospital stay | at patient discharge, an average of 6 days postoperatively
  Days from surgery until discharge.
Maximum voluntary isometric contraction (MVIC) | 24 and 48 hours postoperatively.
  It measures quadriceps strength and is normalized to the body mass index (N * m/kg). This test correlates well with the functional outcome. Will be measured with standard handheld dynamometer (MicroFET2; Hoogan Industries, West Jordan, Utah) perpendicular to the tibial crest 5 cm proximal to the medial malleolus to make the measurement. The patients are told to "reach maximum force and hold for three seconds." Three measurements will be done, and the average will be taken.
  The primary effectiveness endpoints of the study will be the percentage of baselineMVIC retained on the quadriceps of the leg receiving arthroplasty for each subject at 6, 24, and 48 hours postoperatively.
  A higher the percentage will relate with less motor block.

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Biarnes Suñe, M.D., Ph.D., Study Director; Carlos I Salvadores de Arzuaga, M.D., Principal Investigator
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danninger T, Opperer M, Memtsoudis SG. Perioperative pain control after total knee arthroplasty: An evidence based review of the role of peripheral nerve blocks. World J Orthop. 2014 Jul 18;5(3):225-32. doi: 10.5312/wjo.v5.i3.225. eCollection 2014 Jul 18. PMID 25035824
- [Background] Dong CC, Dong SL, He FC. Comparison of Adductor Canal Block and Femoral Nerve Block for Postoperative Pain in Total Knee Arthroplasty: A Systematic Review and Meta-analysis. Medicine (Baltimore). 2016 Mar;95(12):e2983. doi: 10.1097/MD.0000000000002983. PMID 27015172
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Chelly JE, Greger J, Gebhard R, Coupe K, Clyburn TA, Buckle R, Criswell A. Continuous femoral blocks improve recovery and outcome of patients undergoing total knee arthroplasty. J Arthroplasty. 2001 Jun;16(4):436-45. doi: 10.1054/arth.2001.23622. PMID 11402405
- [Background] Sharma S, Iorio R, Specht LM, Davies-Lepie S, Healy WL. Complications of femoral nerve block for total knee arthroplasty. Clin Orthop Relat Res. 2010 Jan;468(1):135-40. doi: 10.1007/s11999-009-1025-1. Epub 2009 Aug 13. PMID 19680735
- [Background] Burckett-St Laurant D, Peng P, Giron Arango L, Niazi AU, Chan VW, Agur A, Perlas A. The Nerves of the Adductor Canal and the Innervation of the Knee: An Anatomic Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):321-7. doi: 10.1097/AAP.0000000000000389. PMID 27015545
- [Background] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- [Background] Elkassabany NM, Antosh S, Ahmed M, Nelson C, Israelite C, Badiola I, Cai LF, Williams R, Hughes C, Mariano ER, Liu J. The Risk of Falls After Total Knee Arthroplasty with the Use of a Femoral Nerve Block Versus an Adductor Canal Block: A Double-Blinded Randomized Controlled Study. Anesth Analg. 2016 May;122(5):1696-703. doi: 10.1213/ANE.0000000000001237. PMID 27007076
- [Background] Wong WY, Bjorn S, Strid JM, Borglum J, Bendtsen TF. Defining the Location of the Adductor Canal Using Ultrasound. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):241-245. doi: 10.1097/AAP.0000000000000539. PMID 28002228
- [Background] Kardash KJ, Noel GP. The SPANK Block: A Selective Sensory, Single-Injection Solution for Posterior Pain After Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Jan-Feb;41(1):118-9. doi: 10.1097/AAP.0000000000000330. No abstract available. PMID 26678763
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346
- [Derived] de Arzuaga CIS, Miguel M, Biarnes A, Garcia M, Naya J, Khoudeir A, Minguell J, Pujol O. Single-injection nerve blocks for total knee arthroplasty: femoral nerve block versus femoral triangle block versus adductor canal block-a randomized controlled double-blinded trial. Arch Orthop Trauma Surg. 2023 Nov;143(11):6763-6771. doi: 10.1007/s00402-023-04960-5. Epub 2023 Jun 30. PMID 37391523